CLINICAL TRIAL: NCT04436705
Title: The Effectiveness of Progressive Muscle Relaxation Technique in Reducing Cancer-related Pain Among Palliative Care Patients: A Randomized Controlled Trial
Brief Title: The Effectiveness of Progressive Muscle Relaxation Technique in Reducing Cancer-related Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Huda Anshasi, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: The University of Jordan
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Cancer-Related Pain
Keywords: Cancer-related pain; Progressive Muscle Relaxation
MeSH Terms: conditions — Cancer Pain | interventions — Autogenic Training; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation (PMR) technique (Experimental): Participants in intervention group continued Progressive Muscle Relaxation (PMR) technique daily for 20 minutes for a total of four weeks addition to usual care. The usual care consists of pharmacological interventions to manage Cancer-related pain.
  Interventions: Other: Progressive Muscle Relaxation (PMR) technique
- control (No Intervention): control group received only usual care for their pain during the study period. The usual care consists of pharmacological interventions to manage Cancer-related pain.

INTERVENTIONS:
Other: Progressive Muscle Relaxation (PMR) technique — The PMR technique utilized in this study was based on the original technique designed by Jacobson (1938) and subsequently modified by Bernstein and Borkovec (1973). The PMR technique involves tensing the individual muscle groups for about 5 seconds for each muscle. Then, allowing them to relax for about 10 seconds, and notice how the muscle feels when it is relaxed in contrast to how it felt when it was tensed. The technique is accompanied by breathing exercises in order to feel the sense of relaxation. In this study, the PMR technique refers to tensing and relaxing the muscles from the forehead to the feet one by one, including the eleven muscle groups (right arm, left arm, forehead, jaw and neck, back and shoulders, stomach, thighs, right calf, left calf, right foot and left foot). The total procedure takes around 20 minutes.
  Arms: Progressive Muscle Relaxation (PMR) technique

SUMMARY:
This randomized controlled trial was designed to evaluate the effectiveness of the Progressive Muscle Relaxation (PMR) technique in reducing Cancer-related Pain (CRP) in patients receiving palliative care in Jordan.

The main hypothesis (H0) of this trial is that cancer patients receiving palliative care do not report a decrease in pain intensity levels and an improve in pain interferences with life activities as a result of participating in PMR technique to a significant extent compared to patients who do not participate. The sub-hypothesis (H1) of this trial is that cancer patients receiving palliative care report a decrease in pain intensity levels and an improve in pain interferences with life activities as a result of participating in PMR technique to a significant extent compared to patients who do not participate.

DETAILED DESCRIPTION:
2. Methods

1. Design:

   This study was designed as an assessor-blinded, prospective, two parallel groups, randomized, controlled trial.
2. Participants and setting:

   Participants were recruited from palliative care outpatient clinics at King Hussein Cancer Center in Amman, Jordan.

   The sample size was calculated using statistical software package G* Power 3.0.10. Based on α = 0.05, a power of 80%, and a medium effect size (Cohen's d = 0.50), the minimum required sample for each group was 64 patients. To be conservative and avoid the negative impact of attrition, the sample was increased to 150 patients for both groups; hence 75 participants were required per group.
3. Randomization:

   The list of potential patients was given weekly to the first author by palliative nurse coordinator. The second author assessed the patients based on study inclusion criteria. A total of fifteen patients were excluded due to not meeting the trial criteria (n=13) and refusing to participate in the trial (n=2). The second author was not engaged in study intervention divided remaining 150 patients into two groups (intervention group (n=75), and control group (n=75)).

   Participants were randomly allocated in a 1:1 ratio to PMR and control groups using a computer-based minimization algorithm stratifying for gender, type of analgesics (non-opioid or weak opioid). The second author informed the participants about the results of randomization by providing labels coded either intervention or control group. Training on PMR technique were done by the first author who was not blinded to study groups. The participants were also not blinded to the study intervention due to the nature of kind of study intervention. All evaluations were completed by a single data collector who was blinded to study groups.

   In this trial, the blinding condition of data collector was maintained by two steps: (1) the first author informed the patients to not provide any information to the data collector about their allocated group, and (2) the data collector reminded all the patients to not reveal what group s/he was randomized to. Thus, the condition of assessor-blind was confirmed in this trial by blinding the data collector. During the study period, one participant in control group due to travel outside the country, and one participant in intervention group due to lack of sufficient time withdrew from the study. Thus, 148 participants completed the study (RMP group (n=74), and control group (n=74)).
4. Procedures:

   The participants received training on the PMR intervention in the palliative care outpatient clinic in a quiet room with adequate light to make them feel relaxed during the intervention. Training on the PMR intervention was delivered individually by face to face. Patients in the intervention group were received instruction on PMR technique by the first author who trained and experienced in the technique. The theoretical session on the PMR took approximately 15 minutes. After the completion of the theoretical session, the first author demonstrated the PMR technique, then the participants applied the technique until they acquired the skill. Participants in intervention group received totally 30 to 40 minutes training on PMR technique including theoretical and practical sessions. Then, PMR booklets designed by the authors were given to the patients in training sessions. Furthermore, the first author recorded PMR technique with a voice recorder using her own voice, and the recorder file was downloaded on compact disc (CD). Each participant was given a copy of the CD to practice PMR technique at home. The intervention group continued the PMR daily for 20 minutes for a total of four weeks at their home. All participants were warned not to take analgesics either orally sixty minutes before or intravenously thirty minutes before the PMR technique. Daily reminder phone calls or Short Message Service (SMS) were performed to remind participants for practicing the technique and check their compliance with study protocol. Regarding to control group, the patients were invited to the same room and completed the baseline assessment. All participants received usual care for their pain during the study period which contained only pharmacological interventions.

   For ethical reasons, after completing this study, the participants in the control group had the opportunity to receive study intervention. These data were not analyzed.
5. Data analysis:

Data were evaluated using Statistical Package for the Social Sciences (SPSS) version 22.0. Patients' demographics, clinical characteristics, and BPI scores were represented as mean values, standard deviations (SD), and percentages. Authors analyzed between-group differences at baseline using t tests for continuous variables and Chi-square tests for categorical variables. The comparisons between two groups in terms of BPI scores were made using Mann-Whitney U test. Additionally, Friedman test was conducted to assess the data for differences in BPI scores within-group. The level of significance was set at p < 0.05 for all tests.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 years and older
* diagnosed with cancer.
* reported complaints of pain ≥1 on a 0-10 Numerical Rating Scale (NRS) in the 24 hours before recruitment.
* were treated with non-opioid or weak opioid analgesic.
* had a Karnofsky Performance Scale Index ≥ 20.
* had regular access to a telephone.

Exclusion Criteria:

* a diagnosis of psychiatric illness, central nervous system tumors and musculoskeletal disorders (because these conditions may limit the effectiveness of PMR technique).
* using any type of complementary therapy during the trial period.
* Patients who had no pain and were treated with strong opioid analgesics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cancer-related pain | The BPI assessment was collected at baseline (T0) ( pre-intervention)
  Brief Pain Inventory (BPI) was used to assess cancer-related pain. The BPI consists of two subscales: (1) pain intensity, and (2) pain interferences with life activities. The pain intensity is evaluated at 4 different times: (1) the worst pain in the last 24 hours, (2) the least pain in the last 24 hours, (3) pain on average, and (4) pain right now. By asking patients to rate their pain on the 0 (no pain) to 10 (pain as bad as you can imagine) rating scale, the average of these 4 items is the person's pain intensity. The second subscale, pain interference, consists of 7 items that evaluate the extent to which pain interferes with general activity, walking, mood, relations with others, working, sleep, and enjoyment of life. Each item is rated on the 0 (does not interfere) to 10 (completely interferes).
Cancer-related pain | The BPI assessment was collected at the end of PMR technique (4 weeks from T0)
  Brief Pain Inventory (BPI) was used to assess cancer-related pain. The BPI consists of two subscales: (1) pain intensity, and (2) pain interferences with life activities. The pain intensity is evaluated at 4 different times: (1) the worst pain in the last 24 hours, (2) the least pain in the last 24 hours, (3) pain on average, and (4) pain right now. By asking patients to rate their pain on the 0 (no pain) to 10 (pain as bad as you can imagine) rating scale, the average of these 4 items is the person's pain intensity. The second subscale, pain interference, consists of 7 items that evaluate the extent to which pain interferes with general activity, walking, mood, relations with others, working, sleep, and enjoyment of life. Each item is rated on the 0 (does not interfere) to 10 (completely interferes).
Cancer-related pain | The BPI assessment was collected at 1-month follow-up (T2)
  Brief Pain Inventory (BPI) was used to assess cancer-related pain. The BPI consists of two subscales: (1) pain intensity, and (2) pain interferences with life activities. The pain intensity is evaluated at 4 different times: (1) the worst pain in the last 24 hours, (2) the least pain in the last 24 hours, (3) pain on average, and (4) pain right now. By asking patients to rate their pain on the 0 (no pain) to 10 (pain as bad as you can imagine) rating scale, the average of these 4 items is the person's pain intensity. The second subscale, pain interference, consists of 7 items that evaluate the extent to which pain interferes with general activity, walking, mood, relations with others, working, sleep, and enjoyment of life. Each item is rated on the 0 (does not interfere) to 10 (completely interferes).

CONTACTS AND LOCATIONS:
Overall Officials: Ministry of Health, Amman, Jordan, Study Director — MOH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anshasi H, Saleh M, Abdalrahim MS, Shamieh O. The effectiveness of progressive muscle relaxation technique in reducing cancer-related pain among palliative care patients: A randomized controlled trial. Br J Pain. 2023 Oct;17(5):501-509. doi: 10.1177/20494637231190191. Epub 2023 Jul 18. PMID 38107755